CLINICAL TRIAL: NCT04447690
Title: Prevalence of Mental Health Problems Among Undergraduate Students at the Universidad de Los Andes
Status: Completed | Type: Observational
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Ministerio de Educación, Chile (Unknown)
Responsible Party: Principal Investigator, Jorge Gaete, Associate Professor, Universidad de los Andes, Chile
Other Study IDs: FDI UAN1901
Record Dates: First submitted 2020-01-24; First posted 2020-06-25 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Student; Mental Health; Depression, Anxiety; Depression; Anxiety; College Drinking; Stress
Keywords: college students; undergraduate
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Alcohol Drinking in College

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project seeks to know the prevalence of mental health problems among undergraduate students, through internationally and nationally validated screening instruments. The project also aims to understand better the associated factors contributing to the mental health problems of this population. Through the critical analysis of the results, our proposal aims to establish the prevalence of anxiety, depression, suicidality and substance use, and the association with socioeconomic features, academic stress, sense of belonging to the university, interpersonal relationships, and sleep habits among other factors. Once finalized the study, the results obtained will be disseminated to the university community and published in peer-reviewed journals.

The results will help the university authorities to design and implement measures to prevent mental health problems in this community.

DETAILED DESCRIPTION:
Background Mental health in the university population has become in recent years a common and serious problem worldwide. There are various studies, systematic reviews and meta-analyses that have been carried out over the past 5 years, which show very worrying figures. In the USA, it has been described in medical students that between 6.0% and 66.5% have depression, between 7.7% and 65.5% anxiety disorders, and between 12.2% and 96.7% refer having stress. In China, on the other hand, a study was reported in 2016 that revealed a prevalence of depression of 23.8%. In Latin America we find a study carried out in Brazil among medical students, which shows a prevalence of depression of 30.6%, anxiety disorders of 32.9, and stress of 49.9%, among other indicators described. In Chile, during 2019 appears the results of the "First National Survey of Mental Health among university students", surveying over 600 students from three universities in Chile. This study showed that 46% of the students presented depressive symptoms, 46% had anxiety symptoms, 53.5% stress symptoms and 29.7% presented all three symptoms simultaneously. In addition, 5.1% of the students reported having suicidal thoughts at the time of the study.

There are multiple determinants that influence mental health, both social, biological, and psychological factors. Within these, the socioeconomic levels of the families of origin and the education attained by their parents stand out, but also the contexts of violence -in its multiple forms- to which university students may be exposed, levels of stress for academic reasons, discrimination for various reasons, in addition to poor health in general.

University students are a group that has certain characteristics in common that makes it particularly vulnerable in terms of their mental health. Among these factors, we can mention: the process of adaptation from the school environment to the university environment, the vocational uncertainty, being subjected to a constant academic workload, responding with demands of both their own and their environment (such as parents and society), and facing worries about entering into the world of work. In short, passing through the university is a period of constant changes, which demands self-management and support, but it also means an adaptation process that can help to eventually develop mental health problems.

At Universidad de los Andes there are no official published figures on the prevalence of mental health problems among university students, nor on possible associated factors among its students. It is important to have a clear and precise current status, as this would allow the implementation of prevention policies, interventions, and the creation of support networks that can help students' mental health.

General Aim:

The general aim of this project is to describe the mental health of the students of the Universidad de los Andes and its association with individual factors, especially academic stress, sense of university belonging, peer violence, substance abuse, and sleep habits.

Methodology Participants. All regular undergraduate students from first to last year of career and older than 18 years old from the Universidad de los Andes will be invited to participate. The various academic units and faculties have offered support and will join the study. Participation is voluntary.

Sample size. Random sampling will be considered for each stratum defined by the career and its year, the sample size is determined from the number of enrolled. For this sample calculation, it has been used as p = 0.1, considering that different studies have estimated the prevalence of suicidal ideation in the last year of 10% (10). A non-response of 20% is anticipated, therfore the sample size is increased by that percentage. A total of 4836 students are expected to participate.

Instruments. A detailed description of the instruments can be found in the Outcomes section of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Regular undergraduate students

Exclusion Criteria:

* Nonconsent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undergraduate regular students of every career from Universidad de los Andes, Chile.
Sampling Method: Non-Probability Sample
Enrollment: 5553 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS-21) | Up to 4 weeks
  Self-reported symptoms with the Depression, Anxiety and Stress Scale (DASS-21), which have 21 items, each scoring between 0 and 3, the minimum score is 0 and the maximum score of 63. The cut-off score for the depression subscale is 6, Anxiety is 5, Stress is 6.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 4 weeks
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire used for suicide assessment. This scale has 6 items and each item has to be answered Yes or No. The total score is 6. A score of 0 is no ideation is present.
CAGE | Up to 4 weeks
  Self-report of harmful alcohol drinking. 4 items. CAGE stands for:
  C: Have you felt the need to Cut down drinking? A: Have you ever felt Annoyed by criticism of drinking? G: Have you had Guilty feelings about drinking? E: Do you ever take a morning Eye opener (a drink first thing in the morning to steady your nerves or get rid of a hangover)? The range score goes from 0 to 4. The point cut off is >= 2.
Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Up to 4 weeks
  Adaptation of The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) interview model, including prescription and nonprescription drugs and vaping. It has 8 items exploring the frequency of substance use in the last 3 months (daily, weekly, yearly) and the problems associated with the use. It explores the use of 10 kinds of drugs.

SECONDARY OUTCOMES:
Sociodemographic characteristics | Up to 4 weeks
  Ad hoc self-report survey:
  * Current age
  * University enrollment year
  * Current years of study
  * Sex
  * Gender
  * Civil status
  * Parenting and number of child(s)
  * Nationality
  * Etnicity
  * Ocupational situation: only study, part-time worker, fulltime worker and study
  * Carrer
  * Maximum parents studies degree: analphabet, school, undergraduate, postgraduate; complete or incomplete studies.
  * Payment of studies: credit, schollarship, self-pay
  * Travel time from home to campus: minutes, hours.
General Health perception | Up to 4 weeks
  Self-perception on a subjective analogous scale of physical health
General Menta Health perception | Up to 4 weeks
  Self-perception on a subjective analogous scale of mental health
History of chronic diseases | Up to 4 weeks
  Ad hoc self-report survey of any previous chronic physical disease
Physical activity | Up to 4 weeks
  Ad hoc self-report survey of minutes of physical activity during the past week
Social activities | Up to 4 weeks
  Ad hoc self-report survey of time spent with friends or social gatherings
Family functionality (APGAR) | Up to 4 weeks
  Family functionality APGAR score: a 5-item measure of perceived family support in the domains of adaptation, partnership, growth, affection, and resolve. E.g. "I find that my family accepts my wishes to take on new activities or make changes in my lifestyle". Scores range from 0 to 10, being 10 a total satisfaction with family functionality.
History of personal and family mental health problems | Up to 4 weeks
  Ad hoc self-report questionnaire of personal and family mental health history:
  * Previous diagnosis of depression, bipolar disorder, panic attacks, anxiety disorders, eating disorders, ADHD.
  * Current psychotherapy of psychiatric medication
  * Family history of psychiatric disorders
Insomnia Severity Index (ISI) | Up to 4 weeks
  Self-report of insomnia perception. it has 7 items, and responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. Scores ranges from 0 to 28. A clinical Insomnia threshold score of 15.
University violence and bullying | Up to 4 weeks
  Ad hoc self-report survey of violence suffered from teachers, administrative, auxiliaries, and other students; discrimination and bullying.
Sexuality and sexual health | Up to 4 weeks
  Ad hoc self-report survey of sexual health, including sexual orientation, the current status of an emotional relationship, number of sex partners in the last year, history of Sexually Transmitted Disease (STD).
Sense of Social and Academic Fit (SSAF) | Up to 4 weeks
  Sense of Social and Academic Fit (SSAF) is a self-report questionnaire of 17 items, with responses on a Likert format from 1-7. It measures academic and social sense of belonging. The score is produced as the average of the scores reported in each item. The minimum score is 1 and the maximum score is 17. A higher score means higher sense of belonging.
COVID-19 questions | Up to 4 weeks
  Ad-hoc self-report survey of current perception and possible diagnosis of COVID-19:
  * Fear or preoccupation about getting COVID-19
  * Sense of severity if diagnosed with COVID-19
  * Fear or preoccupation about a family member or friend to get COVID-19
  * Current diagnosis of COVID-19
  * A family member diagnosed with COVID19
  * Sense of compliance with social isolation and quarantine
  * Persons living with (family, friends, alone)
  * Frequency of: going out of home, gather with others, virtual socialization, keeping a routine, exercise realized, recreative activities, meditation or prayer, seek information about the situation of COVID19
  * Frequency of the following symptoms: nervousness, hopelessness, depression, amount of effort required to realize activities, self-value, anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gaete Olivares, MD, PhD, Study Chair — Universidad de los Andes, Chile
Locations (1):
- Universidad de los Andes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hope V, Henderson M. Medical student depression, anxiety and distress outside North America: a systematic review. Med Educ. 2014 Oct;48(10):963-79. doi: 10.1111/medu.12512. PMID 25200017
- [Background] Lei XY, Xiao LM, Liu YN, Li YM. Prevalence of Depression among Chinese University Students: A Meta-Analysis. PLoS One. 2016 Apr 12;11(4):e0153454. doi: 10.1371/journal.pone.0153454. eCollection 2016. PMID 27070790
- [Background] Stapinski LA, Montgomery AA, Araya R. Anxiety, depression and risk of cannabis use: Examining the internalising pathway to use among Chilean adolescents. Drug Alcohol Depend. 2016 Sep 1;166:109-15. doi: 10.1016/j.drugalcdep.2016.06.032. Epub 2016 Jul 1. PMID 27427415
- [Background] Gobbi G, Atkin T, Zytynski T, Wang S, Askari S, Boruff J, Ware M, Marmorstein N, Cipriani A, Dendukuri N, Mayo N. Association of Cannabis Use in Adolescence and Risk of Depression, Anxiety, and Suicidality in Young Adulthood: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2019 Apr 1;76(4):426-434. doi: 10.1001/jamapsychiatry.2018.4500. PMID 30758486
- [Background] Pigeon WR, Bishop TM, Krueger KM. Insomnia as a Precipitating Factor in New Onset Mental Illness: a Systematic Review of Recent Findings. Curr Psychiatry Rep. 2017 Aug;19(8):44. doi: 10.1007/s11920-017-0802-x. PMID 28616860
- [Background] Taylor DJ, Gardner CE, Bramoweth AD, Williams JM, Roane BM, Grieser EA, Tatum JI. Insomnia and mental health in college students. Behav Sleep Med. 2011;9(2):107-16. doi: 10.1080/15402002.2011.557992. PMID 21491233
- [Background] Hrafnkelsdottir SM, Brychta RJ, Rognvaldsdottir V, Gestsdottir S, Chen KY, Johannsson E, Guethmundsdottir SL, Arngrimsson SA. Less screen time and more frequent vigorous physical activity is associated with lower risk of reporting negative mental health symptoms among Icelandic adolescents. PLoS One. 2018 Apr 26;13(4):e0196286. doi: 10.1371/journal.pone.0196286. eCollection 2018. PMID 29698499
- [Background] Feng Q, Zhang QL, Du Y, Ye YL, He QQ. Associations of physical activity, screen time with depression, anxiety and sleep quality among Chinese college freshmen. PLoS One. 2014 Jun 25;9(6):e100914. doi: 10.1371/journal.pone.0100914. eCollection 2014. PMID 24964250
- [Background] Wu X, Tao S, Zhang Y, Zhang S, Tao F. Low physical activity and high screen time can increase the risks of mental health problems and poor sleep quality among Chinese college students. PLoS One. 2015 Mar 18;10(3):e0119607. doi: 10.1371/journal.pone.0119607. eCollection 2015. PMID 25786030
- [Background] Ploderl M, Tremblay P. Mental health of sexual minorities. A systematic review. Int Rev Psychiatry. 2015;27(5):367-85. doi: 10.3109/09540261.2015.1083949. Epub 2015 Nov 9. PMID 26552495
- [Background] Stojanovic-Tasic M, Grgurevic A, Cvetkovic J, Grgurevic U, Trajkovic G. Association between somatic diseases and symptoms of depression and anxiety among Belgrade University students. Med Glas (Zenica). 2014 Aug;11(2):373-8. PMID 25082256
- [Background] Oswalt SB, Wyatt TJ. Sexual orientation and differences in mental health, stress, and academic performance in a national sample of U.S. college students. J Homosex. 2011;58(9):1255-80. doi: 10.1080/00918369.2011.605738. PMID 21957858
- [Background] Mortier P, Auerbach RP, Alonso J, Bantjes J, Benjet C, Cuijpers P, Ebert DD, Green JG, Hasking P, Nock MK, O'Neill S, Pinder-Amaker S, Sampson NA, Vilagut G, Zaslavsky AM, Bruffaerts R, Kessler RC; WHO WMH-ICS Collaborators. Suicidal Thoughts and Behaviors Among First-Year College Students: Results From the WMH-ICS Project. J Am Acad Child Adolesc Psychiatry. 2018 Apr;57(4):263-273.e1. doi: 10.1016/j.jaac.2018.01.018. Epub 2018 Feb 13. PMID 29588052
- [Background] Bastounis A, Callaghan P, Banerjee A, Michail M. The effectiveness of the Penn Resiliency Programme (PRP) and its adapted versions in reducing depression and anxiety and improving explanatory style: A systematic review and meta-analysis. J Adolesc. 2016 Oct;52:37-48. doi: 10.1016/j.adolescence.2016.07.004. Epub 2016 Aug 2. PMID 27494740
- [Background] Huang J, Nigatu YT, Smail-Crevier R, Zhang X, Wang J. Interventions for common mental health problems among university and college students: A systematic review and meta-analysis of randomized controlled trials. J Psychiatr Res. 2018 Dec;107:1-10. doi: 10.1016/j.jpsychires.2018.09.018. Epub 2018 Sep 29. PMID 30300732
- [Background] Daya Z, Hearn JH. Mindfulness interventions in medical education: A systematic review of their impact on medical student stress, depression, fatigue and burnout. Med Teach. 2018 Feb;40(2):146-153. doi: 10.1080/0142159X.2017.1394999. Epub 2017 Nov 7. PMID 29113526
- [Background] Johnson J, Panagioti M. Interventions to Improve the Breaking of Bad or Difficult News by Physicians, Medical Students, and Interns/Residents: A Systematic Review and Meta-Analysis. Acad Med. 2018 Sep;93(9):1400-1412. doi: 10.1097/ACM.0000000000002308. PMID 29877913
- [Background] Walton GM, Cohen GL. A question of belonging: race, social fit, and achievement. J Pers Soc Psychol. 2007 Jan;92(1):82-96. doi: 10.1037/0022-3514.92.1.82. PMID 17201544
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Fernandez-Mendoza J, Rodriguez-Munoz A, Vela-Bueno A, Olavarrieta-Bernardino S, Calhoun SL, Bixler EO, Vgontzas AN. The Spanish version of the Insomnia Severity Index: a confirmatory factor analysis. Sleep Med. 2012 Feb;13(2):207-10. doi: 10.1016/j.sleep.2011.06.019. Epub 2011 Dec 14. PMID 22172961
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Al-Halabi S, Saiz PA, Buron P, Garrido M, Benabarre A, Jimenez E, Cervilla J, Navarrete MI, Diaz-Mesa EM, Garcia-Alvarez L, Muniz J, Posner K, Oquendo MA, Garcia-Portilla MP, Bobes J. Validation of a Spanish version of the Columbia-Suicide Severity Rating Scale (C-SSRS). Rev Psiquiatr Salud Ment. 2016 Jul-Sep;9(3):134-42. doi: 10.1016/j.rpsm.2016.02.002. Epub 2016 May 2. English, Spanish. PMID 27158026
- [Background] Interian A, Chesin M, Kline A, Miller R, St Hill L, Latorre M, Shcherbakov A, King A, Stanley B. Use of the Columbia-Suicide Severity Rating Scale (C-SSRS) to Classify Suicidal Behaviors. Arch Suicide Res. 2018 Apr-Jun;22(2):278-294. doi: 10.1080/13811118.2017.1334610. Epub 2017 Jul 17. PMID 28598723
- [Background] Saitz R, Lepore MF, Sullivan LM, Amaro H, Samet JH. Alcohol abuse and dependence in Latinos living in the United States: validation of the CAGE (4M) questions. Arch Intern Med. 1999 Apr 12;159(7):718-24. doi: 10.1001/archinte.159.7.718. PMID 10218752
- [Background] Dhalla S, Kopec JA. The CAGE questionnaire for alcohol misuse: a review of reliability and validity studies. Clin Invest Med. 2007;30(1):33-41. doi: 10.25011/cim.v30i1.447. PMID 17716538
- [Background] Ewing JA. Detecting alcoholism. The CAGE questionnaire. JAMA. 1984 Oct 12;252(14):1905-7. doi: 10.1001/jama.252.14.1905. PMID 6471323
- [Background] Bernadt MW, Mumford J, Taylor C, Smith B, Murray RM. Comparison of questionnaire and laboratory tests in the detection of excessive drinking and alcoholism. Lancet. 1982 Feb 6;1(8267):325-8. doi: 10.1016/s0140-6736(82)91579-3. PMID 6120322
- [Background] Knight JR, Sherritt L, Harris SK, Gates EC, Chang G. Validity of brief alcohol screening tests among adolescents: a comparison of the AUDIT, POSIT, CAGE, and CRAFFT. Alcohol Clin Exp Res. 2003 Jan;27(1):67-73. doi: 10.1097/01.ALC.0000046598.59317.3A. PMID 12544008
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- See also: Mental health problems among medical students in Brazil: a systematic review and meta-analysis — http://dx.doi.org/10.1590/1516-4446-2017-2223
- See also: Diagnostic of the prevalence of mental health disorders in college students and associated emotional risk factors — http://dx.doi.org/10.4067/S0717-92272014000300004
- See also: Encuesta Nacional Salud Mental Universitaria — http://www.tvu.cl/prensa/2019/04/29/encuesta-nacional-salud-mental-universitaria-44-de-los-estudiantes-se-han-sometido-a-tratamientos-psicologicos.html
- See also: Bullying and social anxiety experiences in university learning situations — https://doi.org/10.1007/s11218-019-09496-4
- See also: Depression Anxiety Stress Scales (DASS - 21): Validation of the Abbreviated Version in Chilean University Students — https://scielo.conicyt.cl/scielo.php?script=sci_arttext&pid=S0718-48082012000300005
- See also: The depression anxiety stress scale-21: Spanish translation and validation with a Hispanic sample — https://link.springer.com/article/10.1023/A:1016014818163
- See also: Confirmatory Factor Analysis of the Depression-Anxiety-Stress Scales in Depressed and Anxious Patients — https://link.springer.com/article/10.1023/A:1011095624717
- See also: Psychometric Properties of the CAGE Questionnaire for Alcohol Abuse: Results of Three Analyses. — http://www.scielo.org.co/scielo.php?script=sci_abstract&pid=S0034-74502009000200006